CLINICAL TRIAL: NCT00894374
Title: A Single-Dose Bioequivalence Study Comparing Artesunate Tablet (Pfizer) To Arsuamoon® Tablets (Guilin-China) In Healthy Subjects
Brief Title: Bioequivalence Study Comparing Artesunate Tablet To Arsuamoon® Tablets (Guilin-China) In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0551003
Record Dates: First submitted 2009-05-04; First posted 2009-05-07 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Falciparum Malaria
Keywords: Bio-equivalence, Healthy Volunteers
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artesunate (Pfizer) (Experimental)
  Interventions: Drug: Artesunate (Test)
- Artesunate (Arsuamoon® Tablets Guilin-China) (Active Comparator)
  Interventions: Drug: Artesunate (Comparator)

INTERVENTIONS:
Drug: Artesunate (Test) — Oral tablet, single dose, 1 x 100 mg
  Arms: Artesunate (Pfizer)
Drug: Artesunate (Comparator) — Oral tablet, single dose, 2 x 50 mg
  Arms: Artesunate (Arsuamoon® Tablets Guilin-China)

SUMMARY:
The study will determine if artesunate tablet (Pfizer), an antimalarial agent, is pharmaceutically equivalent to Arsuamoon® tablets (Guilin-China).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive.
* BMI of 18 to 30 kg/m2; and a total body weight >45 kg (99 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities.
* A positive urine drug screen, history of regular alcohol consumption.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax of active metabolite of artesunate | 30-Aug-2009

SECONDARY OUTCOMES:
Tolerability | 30-Aug-2009

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0551003&StudyName=Bioequivalence%20Study%20Comparing%20Artesunate%20Tablet%20To%20Arsuamoon%AE%20Tablets%20%28Guilin-China%29%20In%20Healthy%20Subjects